CLINICAL TRIAL: NCT01853046
Title: A Phase I, Multi-center, Non-randomized, Open Label, Parallel-group Study Evaluating the Pharmacokinetics and Safety of Regorafenib (BAY73-4506) in Cancer Subjects With Severe Renal Impairment Compared to a Control Group
Brief Title: Pharmacokinetics and Safety of Regorafenib (BAY73-4506) in Cancer Subjects With Severe Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16653
Record Dates: First submitted 2013-05-10; First posted 2013-05-14 (Estimated); Results first posted 2017-02-20 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2016-12

CONDITIONS: Neoplasms
Keywords: Regorafenib; pharmacokinetics; safety; severe renal impairment; Solid tumors
MeSH Terms: conditions — Neoplasms; Renal Insufficiency | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment (Experimental): Participants with normal/mild renal impairment received Regorafenib 160 mg o.d.as a single dose in Stage 1, Day 1 with a washout of at least 5 days, followed by multiple dosing in an intermittent administration schedule (3 week on / 1 week off) over 2 cycles in Stage 2 (56 days). Cycle 2 started immediately after Cycle 1. A Cycle for this study is defined as 28 days.
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)
- Regorafenib (Stivarga, BAY73-4506)-Severe Renal Impairment (Experimental): Participants with severe renal impairment received Regorafenib 160 mg o.d. as a single dose in Stage 1, Day 1 with a washout of at least 5 days, followed by multiple dosing in an intermittent administration schedule (3 week on / 1 week off) over 2 cycles in Stage 2 (56 days). Cycle 2 started immediately after Cycle 1. A Cycle for this study is defined as 28 days.
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — Regorafenib 160 mg o.d. will be administered as a single dose on Day 1 of Stage 1 followed by multiple dosing in an intermittent administration schedule (3 week-on/1 week-off) over 2 cycles in Stage 2 (56 days, cycle defined as 28 days)

SUMMARY:
To characterize the pharmacokinetics and safety of regorafenib in cancer subjects with severe renal impairment when compared to the Control group (cancer subjects with normal or mildly impaired renal function)

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically confirmed, locally advanced or metastatic, refractory solid tumors who are not candidates for standard therapy
* Male or female subject ≥ 18 years of age
* Women of childbearing potential must have a negative urine pregnancy test performed within 7 days before start of study treatment
* Life expectancy at least 8 weeks
* Adequate bone marrow, and liver function as assessed by the following laboratory requirements conducted within 7 days of starting the study treatment
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2
* For subjects with NORMAL OR MILDLY IMPAIRED RENAL FUNCTION (Control group); to be tested within 7 days of starting the study treatment:

  * Estimated creatinine clearance (CLcr) ≥ 60 mL/min as calculated using the Cockcroft-Gault equation
* For subjects with SEVERELY IMPAIRED renal function; to be tested within 7 days of starting the study treatment:

  * CLcr 15-29 mL/min as calculated using the Cockcroft-Gault equation

Exclusion Criteria:

* Symptomatic metastatic brain or meningeal tumors
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study medication
* History of organ allograft
* Non-healing wound, skin ulcer, or bone fracture
* Pheochromocytoma
* Uncontrolled concurrent medical illness including uncontrolled hypertension
* History of cardiac disease
* Pleural effusion or ascites that causes respiratory compromise
* Interstitial lung disease with ongoing signs and symptoms at the time of screening
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before the start of study medication
* Subjects with evidence or history of bleeding diathesis; any hemorrhage or bleeding event NCI-CTCAE Grade ≥ 3 or higher within 4 weeks of start of investigational treatment
* Dehydration NCI-CTCAEversion 4.0 Grade ≥ 1
* Unresolved toxicity higher than NCI-CTCAE version 4.0 Grade 1 attributed to any prior therapy/procedure (excluding alopecia or anemia or grade 2 neuropathy that is not reversible due to oxaliplatin)
* Seizure disorder requiring anticonvulsant therapy (such as steroids or anti-epileptics)
* For subjects with SEVERELY IMPAIRED renal function:

  * Renal failure requiring hemo- or peritoneal dialysis
  * Acute renal failure
  * Acute nephritis
  * Nephrotic syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-06; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (9):
- United States (5):
  - Los Angeles, California
  - Aurora, Colorado
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - Buffalo, New York
- Canada (4):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 39 adult male or female participants with locally advanced and / or metastatic solid tumors were screened at 4 study centers in Canada and 4 study centers in the USA.
Pre-assignment Details: 15 participants (38.5% of 39) were screening failures and 24 participants received treatment with regorafenib. All 15 participants who failed to meet the inclusion and / or exclusion criteria were not assigned to study
Period: Overall Study
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib (Stivarga, BAY73-4506)-Severe Renal Impairment
Started | 18 | 6
Received Treatment | 18 | 6
Completed | 0 | 0
Not Completed | 18 | 6
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 4 | 2
Not completed — Disease progression | 13 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib (Stivarga, BAY73-4506)-Severe Renal Impairment | Total
Number analyzed (Participants) | 18 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (9.6) | 64.2 (6.9) | 62.5 (8.9)
Gender [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 9 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-tlast) [Area Under the Concentration-time Curve After Single (First) Dose From Time Zero to the Last Data Point >LLOQ (Lower Limit of Quantification)] for Regorafenib and Its Pharmacologically Active Metabolites M-2 and M-5
Description: Based on non-compartmental PK evaluation. The AUC(0-tlast) [Area Under the Concentration-time Curve After Single (First) Dose From Time Zero to the Last Data Point >LLOQ (Lower Limit of Quantification)] is a measure of systemic drug exposure from time 0 up to the time point at which the last measurable drug could be detectable, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Time Frame: Days 1-5: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 24, 48 and 96 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/L
Groups:
- Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment: Participants with severe renal impairment received Regorafenib 160 mg o.d. as a single dose in Stage 1, Day 1 with a washout of at least 5 days, followed by multiple dosing in an intermittent administration schedule (3 week on / 1 week off) over 2 cycles in Stage 2 (56 days). Cycle 2 started immediately after Cycle 1. A Cycle for this study is defined as 28 days.
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 18 | 6
mg*h/L
  Regorafenib | 67.2 (45.5) | 76.6 (50.3)
  Regorafenib metabolites M-2 | 27.8 (80.4) | 19.0 (58.7)
  Regorafenib metabolites M-5 | 5.25 (145) | 2.34 (79.8)
Statistical Analysis 1: Comparison: Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment vs Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment; Point estimates (LS-means) and 2-sided exploratory 90% confidence intervals for AUC(0-tlast) of regorafenib calculated by re-transformation of the logarithmic data from ANOVAs; Test type: Superiority or Other; LS Mean = 1.14, 90% CI 2-sided [0.796 to 1.63]
Statistical Analysis 2: Comparison: Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment vs Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment; Point estimates (LS-means) and 2-sided exploratory 90% confidence intervals for AUC(0-tlast) of metabolites M-2 calculated by re-transformation of the logarithmic data from ANOVAs; Test type: Superiority or Other; LS-means = 0.684, 90% CI 2-sided [0.397 to 1.18]
Statistical Analysis 3: Comparison: Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment vs Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment; Point estimates (LS-means) and 2-sided exploratory 90% confidence intervals for AUC(0-tlast) of metabolites M-5 calculated by re-transformation of the logarithmic data from ANOVAs; Test type: Superiority or Other; LS-means = 0.446, 90% CI 2-sided [0.200 to 0.996]

2. Primary Outcome: AE,ur(0-24) (Amount of Drug Excreted Via Urine During the Collection Interval 0-24 Hours Post Administration) for Metabolites M-7 and M-8
Description: Amount of drug excreted into urine during the collection interval 0-24 hours post dose was expressed as percentage of administered dose.
Time Frame: Days 1-2: 0-24 hours
Population: Participants with a valid pharmacokinetic profile for non compartmental analysis were reported.
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 14 | 5
percentage of dose
  Regorafenib metabolites M-7 | 3.607 (1.124) | 1.309 (0.649)
  Regorafenib metabolites M-8 | 1.120 (0.737) | 0.184 (0.229)

3. Secondary Outcome: AUC (Area Under the Plasma Concentration vs. Time Curve From Zero to Infinity After Single (First) Dose) for Regorafenib and Its Pharmacologically Active Metabolites M-2 and M-5
Description: Based on non-compartmental PK evaluation. AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Time Frame: Days 1-5: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 24, 48 and 96 hours post-dose
Population: Participants with a valid pharmacokinetic profile for non compartmental analysis were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/L
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 18 | 6
mg*h/L
  Regorafenib (n=6, 3) | 59.5 (26.1) | 98.7 (71.0)
  Regorafenib metabolites M-2 (n=13, 4) | 32.6 (89.0) | 20.8 (65.4)
  Regorafenib metabolites M-5 (n=0, 0) | NA (NA) — Number of analyzed subjects is zero. | NA (NA) — Number of analyzed subjects is zero.

4. Secondary Outcome: AUC(0-24) (AUC From Time Zero to 24 Hours p.a. After Single (First) Dose Administration) for Regorafenib and Its Pharmacologically Active Metabolites M-2 and M-5
Description: Based on non-compartmental PK evaluation. The AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample; AUC(0-24) is defined as AUC divided from zero to 24 hours after single (first) dose.
Time Frame: Days 1-5: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10 and 24 hours post-dose
Population: In Normal/mild renal impairment group, participants analyzed for regorafenib, M-2 and M-5 are n=18, 18, and 17 respectively. In Severe renal impairment group, participants analyzed for regorafenib, M-2 and M-5 are n=6, 6, and 5 respectively. Participants with a valid pharmacokinetic profile for non compartmental analysis were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/L
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 18 | 6
mg*h/L
  Regorafenib | 30.0 (39.8) | 28.4 (62.0)
  Regorafenib metabolites M-2 | 13.5 (70.0) | 7.93 (72.7)
  Regorafenib metabolites M-5 | 1.17 (116) | 0.474 (101)

5. Secondary Outcome: Cmax (Maximum Drug Concentration in Plasma After Single (First) Dose Administration) for Regorafenib and Its Pharmacologically Active Metabolites M-2 and M-5
Description: Based on non-compartmental PK evaluation.Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Time Frame: Days 1-5: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 24, 48 and 96 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 18 | 6
mg/L
  Regorafenib | 2.45 (47) | 2.00 (69.7)
  Regorafenib metabolites M-2 | 1.01 (66.7) | 0.525 (69.6)
  Regorafenib metabolites M-5 | 0.0877 (125) | 0.0341 (67.0)

6. Secondary Outcome: Tmax (Time to Reach Maximum Drug Concentration in Plasma After Single (First) Dose) for Regorafenib and Its Pharmacologically Active Metabolites M-2 and M-5
Description: Based on non-compartmental PK evaluation.Tmax refers to the time after dosing when a drug attains its highest measurable concentration (Cmax). It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content.
Time Frame: Days 1-5: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 24, 48 and 96 hours post-dose
Measure: Median (Full Range); unit: h
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 18 | 6
h
  Regorafenib | 4.03 [1.00 to 24.0] | 3.04 [1.00 to 23.75]
  Regorafenib metabolites M-2 | 4.03 [1.00 to 24.0] | 6.04 [1.98 to 23.8]
  Regorafenib metabolites M-5 | 47.8 [6.00 to 96.1] | 48.9 [24.1 to 95.8]

7. Secondary Outcome: Tlast (Time of Last Data Point >LLOQ) After Single (First) Dose for Regorafenib and Its Pharmacologically Active Metabolites M-2 and M-5
Description: based on non-compartmental PK evaluation.
Time Frame: Days 1-5: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 24, 48 and 96 hours post-dose
Measure: Median (Full Range); unit: h
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 18 | 6
h
  Regorafenib | 95.7 [46.4 to 96.3] | 95.8 [95.6 to 96.0]
  Regorafenib metabolites M-2 | 95.7 [46.4 to 96.3] | 95.8 [95.6 to 96.0]
  Regorafenib metabolites M-5 | 95.7 [46.4 to 96.3] | 95.8 [95.6 to 96.0]

8. Secondary Outcome: t1/2 (Half-life Associated With the Terminal Slope) After Single (First) Dose for Regorafenib and Its Pharmacologically Active Metabolites M-2 and M-5
Description: Based on non-compartmental PK evaluation. t1/2 refers to the elimination of the drug. It is the time taken for the blood plasma concentration to reach half the concentration in the terminal phase of elimination. It is expressed in hours (h) and derived from the terminal slope of the concentration versus time curve.
Time Frame: Days 1-5: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 24, 48 and 96 hours post-dose
Population: Participants with a valid pharmacokinetic profile for non compartmental analysis were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 18 | 6
h
  Regorafenib (n=6, 3) | 28.7 (23.0) | 27.9 (32.0)
  Regorafenib metabolites M-2 (n=13, 4) | 26.2 (25.7) | 25.5 (24.0)
  Regorafenib metabolites M-5 (n=0, 0) | NA (NA) — Number of analyzed subjects is zero. | NA (NA) — Number of analyzed subjects is zero.

9. Secondary Outcome: CL/F (Total Body Clearance of Drug After Extravascular Administration) After Single (First) Dose for Regorafenib and Its Pharmacologically Active Metabolites M-2 and M-5
Description: Based on non-compartmental PK evaluation.Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Days 1-5: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 24, 48 and 96 hours post-dose
Population: Participants with a valid pharmacokinetic profile for non compartmental analysis were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/H
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 18 | 6
L/H
  Regorafenib (n=6, 3) | 2.69 (26.1) | 1.62 (71.0)
  Regorafenib metabolites M-2 (n=13, 4) | 5.08 (89.0) | 7.95 (65.4)
  Regorafenib metabolites M-5 (n=0, 0) | NA (NA) — Number of analyzed subjects is zero. | NA (NA) — Number of analyzed subjects is zero.

10. Secondary Outcome: Vz/F (Apparent Volume of Distribution During Terminal Phase After Single (First) Oral Administration) for Regorafenib and Its Pharmacologically Active Metabolites M-2 and M-5
Description: Based on non-compartmental PK evaluation.Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: Days 1-5: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 24, 48 and 96 hours post-dose
Population: Participants with a valid pharmacokinetic profile for non compartmental analysis were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 18 | 6
L
  Regorafenib (n=6, 3) | 111 (31.9) | 65.2 (81.0)
  Regorafenib metabolites M-2 (n=13, 4) | 192 (83.8) | 292 (71.1)
  Regorafenib metabolites M-5 (n=0, 0) | NA (NA) — Number of analyzed subjects is zero. | NA (NA) — Number of analyzed subjects is zero.

11. Secondary Outcome: AUC(0-24)md ((AUC(0-24) After Multiple-dose Administration) for Regorafenib and Its Pharmacologically Active Metabolites M-2 and M-5
Description: Based on non-compartmental PK evaluation.
Time Frame: Days 21-25: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10 and 24 hours post-dose
Population: In Normal/mild renal impairment group, number of participants analyzed is 13. In Severe renal impairment group, number of participants analyzed is 4. Participants with a valid pharmacokinetic profile for non compartmental analysis were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/L
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 18 | 6
mg*h/L
  Regorafenib | 56.0 (56.4) | 45.2 (45.8)
  Regorafenib metabolites M-2 | 53.9 (63.1) | 35.0 (207)
  Regorafenib metabolites M-5 | 49.7 (130) | 34.2 (438)

12. Secondary Outcome: Cmax,md (Cmax After Multiple-dose Administration) for Regorafenib and Its Pharmacologically Active Metabolites M-2 and M-5
Description: as for outcome 5
Time Frame: Days 21-25: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 24, 48 and 96 hours post-dose
Population: Participants with a valid pharmacokinetic profile for non compartmental analysis were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 13 | 4
mg/L
  Regorafenib | 3.52 (54.9) | 2.87 (62.2)
  Regorafenib metabolites M-2 | 3.52 (58.8) | 2.29 (257)
  Regorafenib metabolites M-5 | 3.25 (133) | 2.23 (659)

13. Secondary Outcome: AUC(0-tlast)md (AUC(0-tlast) After Multiple-dose Administration) for Regorafenib and Its Pharmacologically Active Metabolites M-2 and M-5
Description: based on non-compartmental PK evaluation.
Time Frame: Days 21-25: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 24, 48 and 96 hours post-dose
Population: Participants with a valid pharmacokinetic profile for non compartmental analysis were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/L
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 13 | 4
mg*h/L
  Regorafenib | 133 (55.1) | 111 (54.8)
  Regorafenib metabolites M-2 | 136 (64.9) | 92.3 (280)
  Regorafenib metabolites M-5 | 183 (128) | 134 (459)

14. Secondary Outcome: Tmax,md (Time to Reach Maximum Drug Concentration in Plasma After Multiple-dose Administration) for Regorafenib and Its Pharmacologically Active Metabolites M-2 and M-5
Description: based on non-compartmental PK evaluation
Time Frame: Days 21-25: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 24, 48 and 96 hours post-dose
Population: Participants with a valid pharmacokinetic profile for non compartmental analysis were reported.
Measure: Median (Full Range); unit: h
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 13 | 4
h
  Regorafenib | 3.97 [0.000 to 23.8] | 4.25 [0.000 to 10.0]
  Regorafenib metabolites M-2 | 4.12 [0.000 to 23.9] | 4.00 [0.000 to 10.0]
  Regorafenib metabolites M-5 | 0.000 [0.000 to 24.0] | 0.000 [0.000 to 8.00]

15. Secondary Outcome: Tlast,md (Tlast After Multiple-dose Administration) for Regorafenib and Its Pharmacologically Active Metabolites M-2 and M-5
Description: based on non-compartmental PK evaluation
Time Frame: Days 21-25: Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 24, 48 and 96 hours post-dose
Population: Participants with a valid pharmacokinetic profile for non compartmental analysis were reported.
Measure: Median (Full Range); unit: h
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 13 | 4
h
  Regorafenib | 96.0 [48.1 to 96.5] | 95.3 [94.3 to 96.0]
  Regorafenib metabolites M-2 | 96.0 [48.1 to 96.5] | 95.3 [94.3 to 96.0]
  Regorafenib metabolites M-5 | 96.0 [48.1 to 96.5] | 95.3 [94.3 to 96.0]

16. Secondary Outcome: RACmax (Accumulation Ratio Calculated From Cmax,md and Cmax) for Regorafenib and Its Pharmacologically Active Metabolites M-2 and M-5
Description: Based on non-compartmental PK evaluation. Accumulation ratio based on maximum plasma concentration (Cmax) was calculated as ratio of Cmax,md and Cmax.
Time Frame: Up to 25 days
Population: Participants with a valid pharmacokinetic profile for non compartmental analysis were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Accumulation Ratio
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 13 | 4
Accumulation Ratio
  Regorafenib | 1.51 (60.0) | 1.96 (68.2)
  Regorafenib metabolites M-2 | 3.83 (44.9) | 5.94 (216)
  Regorafenib metabolites M-5 | 39.7 (94.0) | 81.8 (515)

17. Secondary Outcome: RAAUC (Accumulation Ratio Calculated From AUC(0-24)md and AUC(0-24)) for Regorafenib and Its Pharmacologically Active Metabolites M-2 and M-5
Description: Based on non-compartmental PK evaluation. RAAUC calculated as ratio of AUC(0-24)md and AUC(0-24).
Time Frame: Up to 25 days
Population: In Normal/mild renal impairment group, participants analyzed for regorafenib, M-2 and M-5 are n=13, 13 and 12 respectively. In Severe renal impairment group, participants analyzed for regorafenib, M-2 and M-5 are n=4, 4 and 3 respectively. Participants with a valid pharmacokinetic profile for non compartmental analysis were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Accumulation Ratio
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 18 | 6
Accumulation Ratio
  Regorafenib | 1.97 (57.1) | 1.96 (52.0)
  Regorafenib metabolites M-2 | 4.32 (45.0) | 6.00 (172)
  Regorafenib metabolites M-5 | 48.3 (76.0) | 87.0 (585)

18. Secondary Outcome: RLin (Linearity Factor Calculated as Ratio From AUC(0-24)md and AUC) for Regorafenib and Its Pharmacologically Active Metabolites M-2 and M-5
Description: Based on non-compartmental PK evaluation. RLin is the linearity factor of PK after multiple administrations of identical doses calculated as ratio of AUC(0-24)md and AUC.
Time Frame: Up to 25 days
Population: Participants with a valid pharmacokinetic profile for non compartmental analysis were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Linearity factor calculated as ratio
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 9 | 2
Linearity factor calculated as ratio
  Regorafenib (n=5, 2) | 0.957 (49.2) | 0.469 (5.24)
  Regorafenib metabolites M-2 (n= 9, 2) | 1.98 (40.7) | 1.19 (144)
  Regorafenib metabolites M-5 (n=0, 0) | NA (NA) — Number of analyzed subjects is zero. | NA (NA) — Number of analyzed subjects is zero.

19. Secondary Outcome: AE,ur(0-24)md (AE,ur(0-24) After Multiple-dose Administration) for Metabolites M-7 and M-8
Description: based on non-compartmental PK evaluation
Time Frame: Days 21-22: 0-24 hours
Population: Participants with a valid pharmacokinetic profile for non compartmental analysis were reported.
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 12 | 4
percentage of dose
  Regorafenib metabolites M-7 | 5.094 (2.322) | 1.647 (0.753)
  Regorafenib metabolites M-8 | 2.566 (1.561) | 1.238 (0.684)

20. Secondary Outcome: AE,ur(0-10) Stage 1 (Amount of Drug Excreted Via Urine During the Collection Interval 0-10 Hours Post Administration) for Metabolites M-7 and M-8
Description: based on non-compartmental PK evaluation
Time Frame: Days 1-2: 0-10 hours
Population: Participants with a valid pharmacokinetic profile for non compartmental analysis were reported.
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 14 | 5
percentage of dose
  Regorafenib metabolites M-7 | 1.752 (0.611) | 0.449 (0.301)
  Regorafenib metabolites M-8 | 0.486 (0.382) | 0.053 (0.089)

21. Secondary Outcome: AE,ur(10-24) Stage 1 ((Amount of Drug Excreted Via Urine During the Collection Interval 10-24 Hours Post Administration) for Metabolites M-7 and M-8
Description: based on non-compartmental PK evaluation
Time Frame: Days 1-2: 10-24 hours
Population: Participants with a valid pharmacokinetic profile for non compartmental analysis were reported.
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 14 | 6
percentage of dose
  Regorafenib metabolites M-7 | 1.855 (0.629) | 0.746 (0.441)
  Regorafenib metabolites M-8 | 0.634 (0.374) | 0.117 (0.133)

22. Secondary Outcome: AE,ur(0-10) Stage 2 for Metabolites M-7 and M-8
Description: based on non-compartmental PK evaluation
Time Frame: Days 21-22: 0-10 hours
Population: Participants with a valid pharmacokinetic profile for non compartmental analysis were reported.
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 12 | 4
percentage of dose
  Regorafenib metabolites M-7 | 2.655 (1.346) | 0.600 (0.255)
  Regorafenib metabolites M-8 | 1.292 (0.902) | 0.469 (0.338)

23. Secondary Outcome: AE,ur(10-24) Stage 2 for Metabolites M-7 and M-8
Description: based on non-compartmental PK evaluation
Time Frame: Days 21-22: 10-24 hours
Population: Participants with a valid pharmacokinetic profile for non compartmental analysis were reported.
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 12 | 4
percentage of dose
  Regorafenib metabolites M-7 | 2.440 (1.098) | 1.047 (0.738)
  Regorafenib metabolites M-8 | 1.274 (0.712) | 0.769 (0.497)

24. Other Pre Specified Outcome: Tumor Response Assessment for Measurable Lesions According to RECIST, v1.1 (Response Evaluation Criteria in Solid Tumors)
Description: Positron emission tomography - computed tomography (ET-CT), CT, or magnetic resonance imaging (MRI) scans of all anatomic regions involved with the disease were performed to assess tumor response using the Response Evaluation Criteria in Solid Tumors, Version 1.1. (RECIST v1.1). Bone metastases were assessed by bone scintigraphy (bone scan). Tumor measurements and evaluation of tumor response were performed at baseline and within the last 7 days of Cycle 2. Thereafter, if subjects continued regorafenib treatment, tumor assessments were performed after every third cycle and at the end-of-treatment (EOT) visit. In addition, outcome of "Assessment of Bone Metastases by Scintigraphy if Applicable (Bone Scan)" was registered, the results of which has been reported as tumor response in this outcome as well.
Time Frame: Up to 6 months
Population: Participants in the Normal/mild renal impairment group had only tumor assessments at screening, thus excluded from efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Renal Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Number analyzed (Participants) | 15 | 6
participants
  Complete response (CR) | 0 | 0
  Partial response (PR) | 0 | 0
  Stable disease (SD) | 10 | 5
  Non CR/Non PD | 0 | 0
  Progressive disease (PD) | 5 | 1
  Not evaluable | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study treatment until 30 days after last dose of study medication.
Description: Safety was assessed routinely and on an ongoing basis
Groups:
- Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Impairment: Participants with normal/mild renal impairment received Regorafenib 160 mg o.d.as a single dose in Stage 1, Day 1 with a washout of at least 5 days, followed by multiple dosing in an intermittent administration schedule (3 week on / 1 week off) over 2 cycles in Stage 2 (56 days). Cycle 2 started immediately after Cycle 1. A Cycle for this study is defined as 28 days.
Arm/Group | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Impairment | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment
Serious Adverse Events (participants affected / at risk) | 9/18 | 2/6
Other Adverse Events (participants affected / at risk) | 18/18 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Impairment (N=18) | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment (N=6)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (3) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (4) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib(Stivarga, BAY73-4506)-Normal/Mild Impairment (N=18) | Regorafenib(Stivarga,BAY73-4506)-Severe Renal Impairment (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 (6) | 2 (5)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (12) | 3 (6)
Abdominal pain lower (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (7) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 8 (16) | 4 (12)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 4 (6) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (3) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (4) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 1 (2)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (20) | 6 (8)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 3 (6) | 2 (8)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (8) | 4 (9)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 3 (3) | 0 (0)
Chills (General disorders) | 2 (2) | 2 (2)
Drug intolerance (General disorders) | 1 (1) | 0 (0)
Early satiety (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 13 (24) | 3 (7)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Medical device site reaction (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 4 (14) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 3 (4) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (2)
Amylase increased (Investigations) | 0 (0) | 1 (8)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (3) | 2 (4)
Blood fibrinogen decreased (Investigations) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (10)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 6 (9) | 1 (3)
Decreased appetite (Metabolism and nutrition disorders) | 11 (23) | 3 (5)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (3) | 1 (1)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (15) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (14) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (6) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (15) | 2 (3)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (5) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2)
Dysgeusia (Nervous system disorders) | 3 (4) | 0 (0)
Headache (Nervous system disorders) | 10 (18) | 2 (5)
Neuropathy peripheral (Nervous system disorders) | 2 (7) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 3 (6)
Urinary retention (Renal and urinary disorders) | 1 (2) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 (12) | 2 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (7) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (7) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 10 (32) | 3 (15)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 5 (12) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 8 (10) | 4 (10)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less